CLINICAL TRIAL: NCT02715024
Title: An Open-label, Randomized, Parallel Study to Evaluate the Clinical Efficacy and Safety of Tamsulosin Alone or in Combination With Solifenacin for the Treatment in Men With Lower Urinary Tract Symptoms Including Overactive Bladder Symptoms
Brief Title: Study to Evaluate the Clinical Efficacy and Safety of Tamsulosin Alone or in Combination With Solifenacin for the Treatment in Men With Lower Urinary Tract Symptoms Including Overactive Bladder Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Taiwan, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAURO-0605-TW
Record Dates: First submitted 2016-03-17; First posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Lower Urinary Tract Symptoms; Overactive Bladder; Benign Prostatic Hyperplasia (BPH)
Keywords: Tamsulosin; Solifenacin; Lower urinary tract symptoms; Overactive bladder
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Bladder, Overactive; Prostatic Hyperplasia | interventions — Tamsulosin; Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tamsulosin alone (Experimental)
  Interventions: Drug: Tamsulosin
- Tamsulosin + solifenacin (Experimental)
  Interventions: Drug: Tamsulosin; Drug: Solifenacin

INTERVENTIONS:
Drug: Tamsulosin — Oral
  Other Names: Harnalidge® D
Drug: Solifenacin — Oral
  Other Names: Vesicare®
  Arms: Tamsulosin + solifenacin

SUMMARY:
The objective of this study is to evaluate the clinical efficacy and safety of tamsulosin alone or in combination with solifenacin for the treatment in men with lower urinary tract symptoms (LUTS) including overactive bladder (OAB) symptoms in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs and symptoms of frequency and urgency related to benign prostatic hyperplasia for at least 3 months
* I-PSS(S) score of ≥ 12
* Maximum flow rate (Qmax) of 4 to15 mL/sec
* Mean urinary frequency of ≥ 8 micturitions per 24 hours and ≥ 1 episode of urgency per 24 hours as verified by the 3-day micturition diary
* Benign digital rectal examination (DRE) result

Exclusion Criteria:

* Clinically significant outflow obstruction
* Significant post void residue volume (PVR >100ml)
* Prostate specific antigen (PSA) ≥10 ng/mL
* Previous or planned prostate surgery, including transurethral resection of the prostate (TURP)
* Transurethral microwave treatment (TUMT), transurethral needle ablation (TUNA), laser, or other invasive or minimally invasive procedures within 12 months
* Patient with a neurological cause for abnormal detrusor activity
* Patients with urinary tract infection, chronic inflammation, bladder stones, bladder neck, sclerosis, urethral stricture, prostatic cancer, severe vesical diverticulum
* Uncontrolled narrow angle glaucoma, urinary or gastric retention or any other medical condition which in the opinion of the investigator makes the use of anticholinergics contra-indicated
* Patients with any other complication which may cause voiding dysfunction
* Patients with severe hepatic dysfunction, severe renal dysfunction, severe cardiovascular disorder, orthostatic hypotension, or senile dementia
* Patients receiving any medication therapy for LUTS/BPH 2 weeks prior to the study
* Use of drugs to treat incontinence currently
* Hypersensitivity to tamsulosin and/or solifenacin or to any component of the formulation
* Any clinically significant condition, which in the opinion of the investigator makes the patients unsuitable for the trial
* Patients had taken any investigational drug in the previous 3 months prior to this study

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2007-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Change in International Prostate Symptoms Score (IPSS-(S)) from baseline to the end of treatment | Baseline and end of treatment (up to 12 weeks)

SECONDARY OUTCOMES:
Change in mean number of urgency episode per 24 hours from baseline to the end of treatment | Baseline and end of treatment (up to 12 weeks)
Change in mean number of micturitions per 24 hours from baseline to the end of treatment | Baseline and end of treatment (up to 12 weeks)
Change in Quality of life index (I-PSS-(L)) from baseline to the end of treatment | Baseline and end of treatment (up to 12 weeks)
Change in maximum flow rate (Qmax) and voided volume determined by uroflowmetry from baseline to the end of treatment | Baseline and end of treatment (up to 12 weeks)
Safety as assessed by adverse events | Up to 12 weeks
Safety as assessed by postvoid residual volume (PVR) | Up to 12 weeks
  Measured by bladder scan
Safety as assessed by vital signs | Up to 12 weeks
Safety as assessed by laboratory parameters | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Therapeutic Area Lead of Medical Affairs (Asia-Oceania), Study Director — Astellas Pharma Taiwan, Inc.
Locations (1):
- Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided